CLINICAL TRIAL: NCT00566774
Title: Myocardial Infarction Free Rx Event and Economic Evaluation (MI FREEE) Trial: a Randomized Evaluation of First-dollar Coverage for Post-MI Secondary Preventive Therapies
Brief Title: A Randomized Evaluation of First-dollar Coverage for Post-MI Secondary Preventive Therapies
Acronym: MI FREEE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Aetna, Inc. (Industry)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor and Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2007-P-000847/1
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: myocardial infarction; secondary prevention; health insurance; cost-sharing
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Full drug coverage
- 2 (Active Comparator)
  Interventions: Other: Usual coverage

INTERVENTIONS:
Other: Full drug coverage — Patients randomized to first-dollar coverage will have their pharmacy benefits changed so that they have no out-of-pocket costs for any beta-blocker, angiotensin converting enzyme inhibitor (ACEI) or angiotensin II receptor blocker (ARB) antagonist, or statin for every subsequent prescription after randomization. All co-pays and co-insurance will be waived at the point of care (i.e. pharmacy) as will any contribution that the cost of these drugs contributes to a patient's deductible
  Arms: 1
Other: Usual coverage — Patients randomized to usual coverage will have no change in their existing benefits
  Arms: 2

SUMMARY:
The objective of this randomized trial is to evaluate the effect of providing full prescription drug coverage (i.e. no co-pays, co-insurance or deductibles) for statins, beta-blockers, angiotensin converting enzyme inhibitors and angiotensin II receptor blockers to patients recently discharged from hospital after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* discharged alive from hospital after acute MI
* receive health services and prescription drug benefits through Aetna, Inc.

Exclusion Criteria:

* enrollment in a Health Savings Account (HSA) plan
* age ≥ 65 years of age at the time of hospital discharge
* plan sponsor has opted out of participating in the study
* receive only medical services or pharmacy coverage but not both through Aetna

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5860 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
First occurrence of fatal or non-fatal acute MI, unstable angina, stroke, congestive heart failure, or revascularization (coronary bypass, stent insertion, or angioplasty) | 2.5 years

SECONDARY OUTCOMES:
First occurrence of fatal or non-fatal acute MI, unstable angina, stroke, or congestive heart failure | 2.5 years
First occurrence of fatal or non-fatal acute MI, unstable angina, stroke, or congestive heart failure or out-of-hospital cardiac death | 2.5 years
Rate of fatal or non-fatal acute MI, unstable angina, stroke, congestive heart failure, or revascularization (coronary bypass, stent insertion, or angioplasty) | 2.5 years
Medication adherence (i.e. the mean medication possession ratio and the proportion of patients fully adherent to each and all 3 of the study medications) | 3 months
Health care utilization (i.e. use of physician visits, emergency room admissions, hospitalizations or other resources) | 3 months
Total pharmacy and health care costs | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- Aetna Inc, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Ito K, Avorn J, Shrank WH, Toscano M, Spettel C, Brennan T, Choudhry NK. Long-term cost-effectiveness of providing full coverage for preventive medications after myocardial infarction. Circ Cardiovasc Qual Outcomes. 2015 May;8(3):252-9. doi: 10.1161/CIRCOUTCOMES.114.001330. Epub 2015 May 5. PMID 25944633
- [Derived] Choudhry NK, Avorn J, Glynn RJ, Antman EM, Schneeweiss S, Toscano M, Reisman L, Fernandes J, Spettell C, Lee JL, Levin R, Brennan T, Shrank WH; Post-Myocardial Infarction Free Rx Event and Economic Evaluation (MI FREEE) Trial. Full coverage for preventive medications after myocardial infarction. N Engl J Med. 2011 Dec 1;365(22):2088-97. doi: 10.1056/NEJMsa1107913. Epub 2011 Nov 14. PMID 22080794
- [Derived] Choudhry NK, Brennan T, Toscano M, Spettell C, Glynn RJ, Rubino M, Schneeweiss S, Brookhart AM, Fernandes J, Mathew S, Christiansen B, Antman EM, Avorn J, Shrank WH. Rationale and design of the Post-MI FREEE trial: a randomized evaluation of first-dollar drug coverage for post-myocardial infarction secondary preventive therapies. Am Heart J. 2008 Jul;156(1):31-6. doi: 10.1016/j.ahj.2008.03.021. Epub 2008 Jun 6. PMID 18585494